CLINICAL TRIAL: NCT03697538
Title: The Effect of Femoral Nerve Block Versus Adductor Canal Block on the Quality of Recovery for Revision Total Knee Arthroplasty, a Prospective Randomized Blinded Study
Brief Title: Adductor Canal Block (ACB) vs Femoral Nerve Block (FNB) in Revision Total Knee Arthroplasty
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Was placed on hold due to the COVID-19 pandemic, and then PI decided not to continue study.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 829859
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Last update posted 2022-09-07 (Actual); Status verified 2022-09

CONDITIONS: Revision Total Knee Arthroplasty
MeSH Terms: interventions — Nerve Block

STUDY DESIGN:
Who Masked: Participant
Masking Description: Patients, nurses on the floor and physical therapists will be blinded to the nature of the patient assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Adductor Canal Block (Experimental): A 20g catheter will be introduced and advanced 2-3 cm beyond the tip of the needle under ultrasound visualization. After needle withdrawal, catheter placement will be checked by visualizing local anesthetic spread under ultrasound. 0.5% ropivacaine will be used for catheter placement. At the conclusion of surgery, the catheters will be connected to a pump that will infuse ropivacaine 0.2% at 6 mL/hr with a patient controlled bolus of 5mL and a lockout of 30 minutes.
  Interventions: Procedure: Nerve Block for pain control post-revision total knee arthroplasty
- Femoral Nerve Block (Active Comparator): A 20g catheter will be introduced and advanced 2-3 cm beyond the tip of the needle under ultrasound visualization. After needle withdrawal, catheter placement will be checked by visualizing local anesthetic spread under ultrasound. 0.5% ropivacaine will be used for catheter placement. At the conclusion of surgery, the catheters will be connected to a pump that will infuse ropivacaine 0.2% at 6 mL/hr with a patient controlled bolus of 5mL and a lockout of 30 minutes.
  Interventions: Procedure: Nerve Block for pain control post-revision total knee arthroplasty

INTERVENTIONS:
Procedure: Nerve Block for pain control post-revision total knee arthroplasty — A 20g catheter will be introduced and advanced 2-3 cm beyond the tip of the needle under ultrasound visualization. After needle withdrawal, catheter placement will be checked by visualizing local anesthetic spread under ultrasound. 0.5% ropivacaine will be used for catheter placement. At the conclusion of surgery, the catheters will be connected to a pump that will infuse ropivacaine 0.2% at 6 mL/hr with a patient controlled bolus of 5mL and a lockout of 30 minutes.

SUMMARY:
This is a prospective, randomized, blinded study with a parallel design and an allocation ratio of 1:1 for the treatment groups. The investigators seek to determine if femoral nerve block (FNB) improves the quality of recovery and improve postoperative analgesia compared with adductor canal block (ACBs) for patients undergoing revision total knee arthroplasty.

DETAILED DESCRIPTION:
This is a prospective, randomized, blinded study with a parallel design and an allocation ratio of 1:1 for the treatment groups. A prospective study design will allow both FNBs and ACBs to be accurately assessed in an effective manner without introducing unnecessary confounding factors. Furthermore, randomization and a parallel design with equal allocation ratio will ensure timely enrollment of patients while also minimizing temporal confounders that may occur with institutional changes to clinical care protocols. Patients, nurses on the floor and physical therapists will be blinded to the nature of the patient assignment (FNB or ACB)

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female patients ages 18-80 scheduled for elective revision TKA.
* American Society of Anesthesiologists (ASA) physical status I -III
* Mentally competent and able to give consent for enrollment in the study.

Exclusion Criteria:

* Patients with any contraindications to regional anesthesia such as infection, nerve injury, anticoagulation.
* Patient refusal.
* Patients with an allergy to local anesthetics or systemic opioids.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2018-10-10 (Actual); Primary Completion 2022-06-27 (Actual); Study Completion 2022-06-27 (Actual)

PRIMARY OUTCOMES:
Quality of recovery-15 item questionnaire (QoR): QoR-15 | 48 hours after surgery
  Our primary objective will be to determine if FNBs will result in improved quality of recovery (QoR-15) compared with ACBs (at 48 hours).
  The questionnaire is 15 questions with a scale from 0-10 on each and composed of two parts; part A and Part B scoring for questions in part A ( questions from 1-10) are scored from 0-10 where 0=none of the time( poor), and 10= all of the time (excellent). Part Bare questions from 11-15 where they are scored from (10-0) where 10=none of the time ( excellent) and 0=all of the time ( poor). The sum of all answers are added together

SECONDARY OUTCOMES:
Opioid consumption | 48 hours post-op
  Opioid requirements during hospitalization will be measured. Total opioid consumption during this time period after surgery will be standardized to morphine equivalent doses and calculated on a milligram basis for this time period or until discharge, whichever occurs first
Pain score measurement: we will use Numeric rating scale for measurement (NRS) | 48 hours post-op
  Pain scores on a 0-10 numerical rating scale (NRS) where 0= no pain and 10= the worst pain ever. the scores will be assessed every 8 hours from nursing documentation through 48 hours or until discharge, whichever occurs first

CONTACTS AND LOCATIONS:
Overall Officials: Nabil M Elkassabany, MD, MSCE, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No